CLINICAL TRIAL: NCT01946490
Title: Time Trends in Diagnostic Delay and Waiting Times of Four Patient Cohorts, Diagnosed With Non-small Cell Lung Cancer, Treated With High Dose Radiotherapy.
Brief Title: Time Trends in Waiting Times of NSCLC Patients.
Status: Withdrawn | Type: Observational
Why Stopped: Not subsidized, will not start in the near future
Sponsor: Maastricht Radiation Oncology (Other)
Collaborators: Comprehensive Cancer Centre The Netherlands (Other)
Responsible Party: Sponsor
Other Study IDs: Waiting Times
Record Dates: First submitted 2013-09-03; First posted 2013-09-19 (Estimated); Last update posted 2015-09-30 (Estimated); Status verified 2015-09

CONDITIONS: Non-Small Cell Lung Cancer
MeSH Terms: conditions — Carcinoma, Non-Small-Cell Lung

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (4):
- Radiotherapy in 2001
- Radiotherapy in 2004
- Radiotherapy in 2006
- Radiotherapy in 2010

SUMMARY:
A large group of non-small cell lung cancer patients is treated with radiotherapy. Delivery of very high radiation doses is needed to obtain local control, but due to the large tumor and nodal volume this is often impossible without causing unrepairable damage to the normal tissue of the mediastinum, spinal cord, esophagus and lung.

Although every tumor is different with respect to the speed with which it grows and spreads, it is obvious that time plays an important role in cancer therapy. Recently it was reported that disease progression or increase of tumor volume occurred during the time interval between diagnosis and treatment.(1, 2) This could lead to a less optimal radiation treatment and consequently have an impact on overall survival. Moreover, the increasing number of diagnostic procedures, aimed at obtaining more accurate information about the tumor extension and biology, as well as the use of more sophisticated but labor intense radiation techniques could prolong the time interval between clinical symptoms and the start of the treatment. However, the influence of new diagnostic procedures or the applied radiotherapy techniques on waiting times is not yet known. The investigators therefore want to investigate 1) time trends in the waiting time for NSCLC patients, 2) the correlation between waiting times and the use of more advanced diagnostic or therapeutic procedures, and 3) the correlation between waiting times and overall survival.

The hypotheses of the study:

1. The diagnostic delay for NSCLC patients has increased during the last 12 years.
2. The preparation time for radiotherapy of NSCLC patients has increased during the last 12 years.
3. Prolonged waiting times are associated with worse overall survival outcome.

DETAILED DESCRIPTION:
A large group of non-small cell lung cancer patients is treated with radiotherapy. Delivery of very high radiation doses is needed to obtain local control, but due to the large tumor and nodal volume this is often impossible without causing unrepairable damage to the normal tissue of the mediastinum, spinal cord, esophagus and lung.

Although every tumor is different with respect to the speed with which it grows and spreads, it is obvious that time plays an important role in cancer therapy. Recently it was reported that disease progression or increase of tumor volume occurred during the time interval between diagnosis and treatment.(1, 2) This could lead to a less optimal radiation treatment and consequently have an impact on overall survival. Moreover, the increasing number of diagnostic procedures, aimed at obtaining more accurate information about the tumor extension and biology, as well as the use of more sophisticated but labor intense radiation techniques could prolong the time interval between clinical symptoms and the start of the treatment. However, the influence of new diagnostic procedures or the applied radiotherapy techniques on waiting times is not yet known. The investigators therefore want to investigate 1) time trends in the waiting time for NSCLC patients, 2) the correlation between waiting times and the use of more advanced diagnostic or therapeutic procedures, and 3) the correlation between waiting times and overall survival.

The hypotheses of the study:

1. The diagnostic delay for NSCLC patients has increased during the last 12 years.
2. The preparation time for radiotherapy of NSCLC patients has increased during the last 12 years.
3. Prolonged waiting times are associated with worse overall survival outcome.

The IKL collected data on waiting times and treatment of NSCLC patients treated in 2001 and 2004. These data will be used for this project. In addition, the MAASTRO lung database contains information of patients treated in 2006 and 2010. Additional information about the diagnostic procedure and radiation treatment preparation will be collected by reviewing the patient charts. For this study a data request has to be submitted to the IKL and access to MAASTRO patient data (charts and EMD) is needed.

The investigators aim to collect the following variables: Date of consultation pulmonologist; Date of multidisciplinary meeting; Date of first consultancy at radiotherapy; Date of start radiotherapy; Information about diagnostic procedure (PET/CT/Pathology/EBUS/EUS); Information about RT procedure (3Dconventional/IMRT); General patient characteristics; Overall survival

ELIGIBILITY:
Inclusion Criteria:

Patients with NSCLC treated in the Dutch province Limburg from 2001 onwards.

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Four cohorts of NSCLC patients will be analyzed. Patients were all treated with radiotherapy with or without chemotherapy. To investigate the time trends, cohorts referred for radiotherapy treatment in 2001, 2004, 2006 and 2010 will be analyzed.
Sampling Method: Non-Probability Sample
Enrollment: 0 (Actual)
Dates: Start 2015-12; Primary Completion 2016-09 (Estimated); Study Completion 2016-09 (Estimated)

PRIMARY OUTCOMES:
Analysis of waiting times | From intake to start of radiotherapy
  Retrospective analysis of the time passed between consultation and start of radiotherapy (an expected average time frame of two weeks).
Correlation of waiting times and treatment outcome | From treatment until date of censoring (12 years)
  Is there a correlation between the time passed between consultation and start of radiotherapy and treatment outcome? (Time frame: 12 years)

CONTACTS AND LOCATIONS:
Locations (1):
- MAASTRO clinic, Maastricht, Limburg, Netherlands